CLINICAL TRIAL: NCT04156568
Title: A Multicentre, Cohort Study of Screening and Preventive Intervention for Latent Tuberculosis Infection in Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Adong Shen, Deputy Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCH_LTBI study 001
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Children LTBI
Keywords: Children; LTBI; Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6INH Group (Experimental): 10mg/kg 6INH were used in this group.
  Interventions: Drug: INH、RFT
- 3INH+RFT group (Experimental): 3INH+RFTwere used in this grroup.
  Interventions: Drug: INH、RFT

INTERVENTIONS:
Drug: INH、RFT — 6INH 10mg/kg 3INH+RFT 15mg/kg

SUMMARY:
The management of latent Mycobacterium tuberculosis infection is a new priority action for the WHO End Tuberculosis (TB) Strategy. However, national guidelines on latent tuberculosis infection testing and treatment have not yet been developed in children of China. Here, we present the results from the 3-year follow-up of a study that aimed to track the development of active disease in individuals with latent tuberculosis infection, identify priority populations for latent infection management, and explore the most suitable latent infection diagnostic approach.

DETAILED DESCRIPTION:
1. Baseline analysis of a population-based, multicentre, prospective cohort study

1. A baseline survey of a population-based, multicentre, prospective cohort study were took in children (≤18).
2. Eligible participants were identifi ed by door-to-door survey with a household sampling design.
3. Participants were screened for active tuberculosis and history of tuberculosis then used a tuberculin skin test and an interferon-γ release assay (QuantiFERON [QFT]) to test for latent infection.

2. Incidence of active tuberculosis in individuals with latent tuberculosis infection in children of China under different treatment regimens

1. Individuals who had tuberculosis infection at baseline (QFT-positivity or TST tuberculin reaction size [induration] of ≥10 mm) were divided and treatment with different therapeutic schedule.
2. Follow-up study were conducted to assess the proportion of latent TB infection converted to active TB

ELIGIBILITY:
Inclusion Criteria:

* Children (0-18 years old).
* Children with QFT-positive or TST induration ≥10 mm).

Exclusion Criteria:

* Patients are allergic to anti-tuberculsis drugs.
* Parents and/or guardians do not agree to participate in this study.
* Participants with active tuberculosis.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity | During the 2 year follow-up study
  Percentage of latent TB infections converted to active TB
Proportion of adverse reactions | During the 2 year follow-up study
  The incidence of adverse reactions in different treatment regimens
Proportion of lost to follow-up | During the 2 year follow-up study
  The proportion of lost to follow-up in different treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: A-Dong Shen, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, China